CLINICAL TRIAL: NCT05259748
Title: The Effect of Psychoeducation Based on the Transtheoretical Model on Healthy Lifestyle Behaviors in Individuals With Schizophrenia: Randomized Controlled Trial
Brief Title: The Effect of Psychoeducation on Healthy Lifestyle Behaviors in Individuals With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatay Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sercan Mansuroglu, Principal Investigator, Hatay Training and Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10378149
Record Dates: First submitted 2021-11-29; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Transtheoretical Model; Healthy Lifestyle; Behavioral Change; Mental Health and Psychiatric Nurse
MeSH Terms: conditions — Schizophrenia; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is conducted in pretest-posttest randomized controlled experimental research type.
Who Masked: Participant
Masking Description: The control group included in the study was not informed about the planned interventions to the experimental group before the study. Necessary information about the intervention study performed on the experimental group was given to the control group after the study was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): At the beginning, personal information form, behavioural change stage diagnosis form and healthy lifestyle scale II were applied. 6-week psychoeducation, consisting of 6 modules, based on the Transtheoretical model, was applied to the intervention group. Finally, posttests were applied after the psychoeducation.
  Interventions: Behavioral: Psychoeducation Based on the Transtheoretical Model on Healthy Lifestyle Behaviors
- control group (No Intervention): At the beginning, personal information form, behavioural change stage diagnosis form and healthy lifestyle scale II were applied. No interventions were applied to the control group. It was contacted with the control group three times, two face to face and one via phone. In the third and final meeting, when the intervention group's sessions are completed, posttests were applied again to the control group.

INTERVENTIONS:
Behavioral: Psychoeducation Based on the Transtheoretical Model on Healthy Lifestyle Behaviors — Healthy lifestyle behaviours psychoeducation programme, based on the Transtheoretical Model, with 6 sessions (healthcare responsibility, nutrition, physical activity, spiritual development, interpersonal relationships, stress management) was applied to the intervention group for 6 weeks as three days in the weekdays and two sessions in a day. Psychoeducation was carried out by the researcher on the same day but within different time zones. Each psychoeducation session took 90-120 minutes with the breaks taken considering the participants' mood. After completing six sessions, the behavioural change identification form and Healthy Lifestyle Behaviors Scale II were applied to the intervention group again.
  Arms: intervention group

SUMMARY:
Definition: Schizophrenia is a chronic mental disorder that causes drastic changes in life quality and life functions, characterized by behavioural, cognitive and affective state deterioration. Therefore, it is regarded as one of the most important health problems causing both personal and economic problems around the world. Unhealthy lifestyle behaviours in individuals with chronic mental disorders, like schizophrenia, are emphasized to play a big part in physical health problems. For individuals to develop a healthy lifestyle behaviour, it is necessary to primarily determine the lifestyle behaviours and then prevent the illnesses caused by the lifestyle and deaths linked to these illnesses. Current theory or models used to benefit from health programmes, prepared for the development of healthy lifestyle behaviours, should be deep-scaled. Theories and models are guides for systematic planning and decision-making. A well-defined model could contribute to the process of effective health improvement programmes for directive and content creation. One of the models mainly used to develop a behavioural change in health and explain how to obtain the most effective health behavioural change is the "Transtheoretical Model". Objective: The study was conducted with the pretest-posttest randomized controlled trial design to detect the effect of psychoeducation on a healthy lifestyle, based on the Transtheoretical Model in an individual with schizophrenia.

The Hypotheses of the Study Hypothesis 1: When the individuals with schizophrenia who received psychoeducation based on the Transtheoretical Model are compared to the ones that did not, they will show progress in behavioural change steps.

Hypothesis 2: When the individuals with schizophrenia who received psychoeducation based on the Transtheoretical Model are compared to the ones that did not, they will have higher final test results in the healthy lifestyle scale.

Methods: The data were collected from 82 participants, as 41 intervention and 41 control. The data were collected via personal information form, behavioural change stage diagnosis form and healthy lifestyle scale II. 6-week psychoeducation, consisting of 6 modules, based on the Transtheoretical model, was applied to the intervention group. No interventions were applied to the control group. Pretests and posttests were applied to both groups.

DETAILED DESCRIPTION:
This study is conducted in pretest-posttest randomized controlled experimental research type in a Community Mental Health Center in the south of Turkey. The population of the study are the individuals with schizophrenia who registered in a Community Mental Health Center and are under observation (N=230). The sample number is determined based on another similar study with power analysis. In the evaluation completed according to the healthy lifestyle behaviours score, the sample number needed to participate in the study was determined to be at least 42 (intervention group=21 - control group=21) in order for research results to have a meaningful effect.In order to reduce the selection bias in the determination of intervention and control groups, intervention and control groups were formed with a third person who did not have a direct role in the research from 1 to 82 using simple random sampling method. The data were collected from 82 individuals with schizophrenia, as 41 intervention and 41 control groups. The individuals with schizophrenia in the study and their families were informed according to the Helsinki Declaration and written and verbal approval were collected. The behavioural change identification form was applied to individuals with schizophrenia, who agreed to participate in the study, and their stage of the Transtheoretical Model was detected. The participants meeting the criteria in the participation stage (contemplation, preparation, action) were assigned to the intervention and control groups with the randomization. Pretests (personal information form, behavioural change identification form, Healthy Lifestyle Behaviours Scale II) were applied to the intervention and control groups before the psychoeducation. In addition to the rehabilitation activities conducted in the Community Mental Health Center, healthy lifestyle behaviours psychoeducation programme, based on the Transtheoretical Model, with 6 sessions (healthcare responsibility, nutrition, physical activity, spiritual development, interpersonal relationships, stress management) was applied to the intervention group for 6 weeks as three days in the weekdays and two sessions in a day. Psychoeducation was carried out by the researcher on the same day but within different time zones. Each psychoeducation session took 90-120 minutes with the breaks taken considering the participants' mood. After completing six sessions, the behavioural change identification form and Healthy Lifestyle Behaviours Scale II were applied to the intervention group again. On the other hand, the control group continued their rehabilitation practices prepared for themselves in the Community Mental Health Center. It was contacted with the control group three times, two face to face and one via phone. In the third and final meeting, when the intervention group's sessions are completed, the behavioural change identification form and Healthy Lifestyle Behaviours Scale II were applied again to the control group. All the participants remained in the study at the end of it. The study was completed with 41 individuals in the intervention group and 41 individuals in the control group. Statistical Package for the Social Sciences v23.0, which is a statistical analysis programme, was used to evaluate the findings of the study. It was benefited from descriptive statistics such as frequency, percentage, arithmetic average, standard deviation, minimum and maximum during data analysis. Parametric tests were used for the data analysis. The chi-squared test was used for relation analysis of two different categorized variables whereas the t-test was used while comparing averages of two independent groups. To determine the alteration of individuals' behavioural change stages before and after receiving psychoeducation, the McNemar test was used. Analysis of covariance (ANCOVA) while detecting the effect of the intervention study in the researches designed in the entrepreneurial pattern. In ANCOVA, to detect how big the effect of the independent variable on the dependent variable the eta squared (effect size) was calculated and the eta squared value (η2) was interpreted that it presents which parts of the change explain the total variant that the independent variable has on the dependent variable and it received a value. Eta squared is interpreted as 0,01 as the minor effect, 0,06 as medium effect and 0,14 as large effect. All test results were evaluated in terms of p<0.05 meaningfulness level

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 18 and 65
* Being diagnosed with schizophrenia according to The Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V)
* Being literate
* Not having education and language problem that can block the interview
* Being open to communication and cooperation
* Being in one of the three stages of the Transtheoretical Model: contemplation, preparation and action

Exclusion Criteria:

* Those who did not meet the inclusion criteria were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Change in the Behavioural Change Stage Identification Form | It was applied as a pre-test before the intervention and as a post-test 6 weeks after the intervention, within 1 week, and the change was observed.
  It was constructed by the researcher using the behavioral change stages of the transtheoretic model and to determine the behavioral stages of the participants in the areas of taking responsibility for their own health, nutrition, physical exercise, spiritual development, stress management and interpersonal relationships.. The structure of the model consists of stages as pre-contemplation, contemplation, preparation, action, maintenance and termination. These stages also describe the individuals' intention, attitude and behavioral change time, as well as their interests and motivations for change. The purpose of using this form is to determine which change stage the participants are in. Thus, it was aimed to provide each individual with the support they need at the stage they are in, to develop and to determine the effectiveness of the psychoeducation given by applying this form before and after the intervention.
Healthy Lifestyle Behaviours Scale-change in health responsibility sub-dimension | It was applied as a pre-test before the intervention and as a post-test 6 weeks after the intervention, within 1 week, and the change was observed.
  Health responsibility is an individual's active sense of responsibility for their own well-being. It is to take care of his own health, to be informed about health, to seek professional help when necessary. With this subscale of the healthy lifestyle behaviors scale, it was aimed to determine the health responsibility levels of the participants. With the psychoeducation planned for 6 weeks, it was aimed to determine and compare the health responsibility levels of the participants before and after the intervention and to evaluate the effectiveness of the intervention.
Healthy Lifestyle Behaviours Scale-change in physical exercise sub-dimension | It was applied as a pre-test before the intervention and as a post-test 6 weeks after the intervention, within 1 week, and the change was observed.
  Physical exercise includes regular practice of light, moderate and heavy exercises. It is carried out in a planned way as a part of daily life. With this subscale of the healthy lifestyle behaviors scale, it was aimed to determine the physical exercise levels of the participants. With the psychoeducation planned for 6 weeks, it was aimed to determine and compare the physical exercise levels of the participants before and after the intervention and to evaluate the effectiveness of the intervention.
Healthy Lifestyle Behaviours Scale-change in nutrition sub-dimension | It was applied as a pre-test before the intervention and as a post-test 6 weeks after the intervention, within 1 week, and the change was observed.
  Nutrition determines the value of an individual in choosing, arranging and choosing meals. With this sub-scale of the healthy lifestyle behaviors scale, it was aimed to determine the nutrition levels of the participants. With the psychoeducation planned for 6 weeks, it was aimed to determine and compare the nutritional levels of the participants before and after the intervention and to evaluate the effectiveness of the intervention.
Healthy Lifestyle Behaviours Scale-change in spiritual development sub-dimension | It was applied as a pre-test before the intervention and as a post-test 6 weeks after the intervention, within 1 week, and the change was observed.
  Spiritual development focuses on the development of inner resources. Growth can happen by relating and being transcended. Transcending provides inner peace, creating the possibility of providing opportunities for more new experiences outside of who we are and what we do. To relate is to be in relationship with the universe and to feel in harmony. Growth is working for life's purposes, maximizing the individual's power towards well-being. With this sub-scale of the healthy lifestyle behaviors scale, it is aimed to determine the spiritual development levels of the participants. With the psychoeducation planned for 6 weeks, it was aimed to determine and compare the spiritual development levels of the participants before and after the intervention and to evaluate the effectiveness of the intervention.
Healthy Lifestyle Behaviours Scale-change in interpersonal relationships sub-dimension | It was applied as a pre-test before the intervention and as a post-test 6 weeks after the intervention, within 1 week, and the change was observed.
  Interpersonal relationships are relationships with others, requiring using communication to establish a meaningful relationship outside of causal requirements. Communication involves sharing thoughts and feelings through verbal and non-verbal messages. With this subscale of the healthy lifestyle behaviors scale, it was aimed to determine the interpersonal relationship levels of the participants. With the psychoeducation planned for 6 weeks, it was aimed to determine and compare the interpersonal relationship levels of the participants before and after the intervention and to evaluate the effectiveness of the intervention.
Healthy Lifestyle Behaviours Scale- change in stress management sub-dimension | It was applied as a pre-test before the intervention and as a post-test 6 weeks after the intervention, within 1 week, and the change was observed.
  Stress management is the individual's ability to identify and activate physiological and psychological resources in order to reduce or effectively control tension. With this subscale of the healthy lifestyle behaviors scale, it was aimed to determine the stress management levels of the participants. With the psychoeducation planned for 6 weeks, it was aimed to determine and compare the stress management levels of the participants before and after the intervention and to evaluate the effectiveness of the intervention.
change in total of the Healthy Lifestyle Behaviours Scale points | It was applied as a pre-test before the intervention and as a post-test 6 weeks after the intervention, within 1 week, and the change was observed.
  The scale measures behaviors that develop health in relation to the healthy lifestyle of the individual. The scale has a total of 52 items and has 6 sub-factors. The subgroups are spiritual development, health responsibility, physical activity, nutrition, interpersonal relations and stress management. The general score of the scale provides a healthy lifestyle behavior score. The lowest score 52 for the entire scale is 52, the highest score is 208.It was aimed to compare and evaluate the efficacy of the healthy lifestyle behavior of the participants before and after the planned psychoeducation as 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sercan Mansuroğlu, Dr., Principal Investigator — Hatay Training and Research Hospital
Locations (1):
- Antakya Community Mental Health Center, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Derived] Mansuroglu S, Kutlu FY. The Transtheoretical Model based psychoeducation's effect on healthy lifestyle behaviours in schizophrenia: A randomized controlled trial. Arch Psychiatr Nurs. 2022 Dec;41:51-61. doi: 10.1016/j.apnu.2022.07.018. Epub 2022 Jul 20. PMID 36428075

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT05259748/Prot_SAP_000.pdf